CLINICAL TRIAL: NCT03515590
Title: Impact of Emulsion Droplet Physical State on Postprandial Lipemia and Satiety in Healthy Adults
Brief Title: Emulsion Droplet Physical State on Postprandial Lipemia and Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Amanda Wright, Ph.D., Associate Professor, University of Guelph
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 1801005
Record Dates: First submitted 2018-04-11; First posted 2018-05-03 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Postprandial Lipemia; Satiety
MeSH Terms: interventions — Emulsions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emulsion with solid droplets (Experimental): Emulsion with solid droplets will be consumed by participants in one study visit along with 1500 mg of crushed and dissolved acetaminophen.
  Interventions: Other: Emulsion with solid droplets
- Emulsion with liquid droplets (Experimental): Emulsion with liquid droplets will be consumed by participants in one study visit along with 1500 mg of crushed and dissolved acetaminophen.
  Interventions: Other: Emulsion with liquid droplets

INTERVENTIONS:
Other: Emulsion with solid droplets — This will be a 500 mL beverage emulsion in which the droplets are crystalline. It will have identical composition to the other intervention, i.e. in one the lipid droplets are solid (i.e. crystallized) and the other in which they remain liquid will be introduced at least 7 days apart. The differences in physical state will be achieved simply by changing the temperatures the emulsions are held at. The emulsion will contain 10 % of the lipid palm stearin with 0.4% of the emulsifier sorbitan monostearate (Span60).
  Arms: Emulsion with solid droplets
Other: Emulsion with liquid droplets — This will be a 500 mL beverage emulsion in which the droplets are liquid. It will have identical composition to the other intervention, i.e. in one the lipid droplets are solid (i.e. crystallized) and the other in which they remain liquid will be introduced at least 7 days apart. The differences in physical state will be achieved simply by changing the temperatures the emulsions are held at. The emulsion will contain 10 % of the lipid palm stearin with 0.4% of the emulsifier sorbitan monostearate (Span60).
  Arms: Emulsion with liquid droplets

SUMMARY:
The purpose of this study is to compare the changes in blood lipids and feelings of satiety after consumption of oil-in-water emulsions in which the droplets are in either the liquid or solid (i.e. crystalline) states.

DETAILED DESCRIPTION:
A double blinded randomized cross-over acute meal study will be carried out in which 15 healthy male participants will attend two study visits, separated by at least one week. On each study visit, fasted participants will consume either the solid or the liquid emulsion, in a randomized order. Both emulsions tested will have the exact same composition only differing in the physical state of the lipid emulsions, in order to isolate the impact of physical state, specifically, on metabolic response. Postprandial lipemia and satiety will be measured for 6 hours after consumption of the test beverage. The study meals will include crushed acetominophen, the appearance of which will be measured in plasma as a measure of liquid content gastric emptying. Participants will be asked to maintain their usual lifestyle habits throughout the study, with some changes in the 48 hour period leading up to each of the two visits.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 18 - 26 kg/m2
* generally healthy
* non-smoking
* non to moderate alcohol drinkers
* fasting plasma cholesterol level <5.2 mmol/L
* plasma triacylglycerol level <1.7 mmol/L
* plasma glucose level <5.6 mmol/L

Exclusion Criteria:

* History of major medical conditions
* taking prescription medications/ over the counter medications
* taking natural health products/ dietary supplements (other than a multivitamin)
* oral antibiotic use in the previous 3 months
* planning to take oral antibiotics in the next 3 months
* food allergy/anaphylactic/life-threatening allergy
* smokers/ regular users of recreational drugs
* elite/ training athletes
* significant weight loss/ gain during the past 3 months
* previous reaction/ sensitivity to acetaminophen
* inability to avoid taking acetaminophen for 48 hours
* sensitivity to the artificial sweetener Sugar Twin® Sucralose and artificial vanilla extract
* not willing to consume Sugar Twin® Sucralose or Artificial vanilla.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Triacylglycerols | 6 hours
  Fasting and postprandial blood sample analysis

SECONDARY OUTCOMES:
Satiety ratings | 6 hours
  Visual analogue scale ratings of feelings of hunger, fullness, appetite, fatigue, after consuming the emulsion beverage. 0: not hungry, empty, no appetite and no fatigue and 10: very hungry, very full, can eat a lot and very fatigued. The distance from the left end of the scale will be measured.
Gastric emptying | 6 hours
  The rate of appearance of acetaminophen (consumed crushed in water immediately after test meal) in the plasma will be determined.
Cholecystokinin | 6 hours
  Fasting and postprandial blood sample analysis
Fatty acid composition | 6 hours
  Fasting and postprandial blood sample analysis
Apolipoprotein B48 | 6 hours
  Fasting and postprandial blood sample analysis
Chylomicron size | 6 hours
  Fasting and postprandial blood sample analysis

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Wright, PhD, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

REFERENCES:
- [Derived] Thilakarathna SH, Hamad S, Cuncins A, Brown M, Wright AJ. Emulsion Droplet Crystallinity Attenuates Postprandial Plasma Triacylglycerol Responses in Healthy Men: A Randomized Double-Blind Crossover Acute Meal Study. J Nutr. 2020 Jan 1;150(1):64-72. doi: 10.1093/jn/nxz207. PMID 31495898